Cover page

May 1, 2016

NCT number NCT03171688

Official Title: Risk Factors for Nausea and Vomiting After Cesarean

Internal study ID: NVPOCesarianasGabriel2017

## Study protocol

- 1. Eligible patients will be invited to participate when cesarean section is indicated and the anesthesiologist asked to provide anesthesia.
- 2. We will begin the informed consent protocol.
- 3. Specific data will be collected before operating room: identification, age, previous PONV status (no previous surgery, previous surgery and no PONV, previous surgery and ponv), history of motion sickness, gestational age, smoking status, nausea in the first trimester, nausea in the third trimester.
- 4. More data will be collected in the operating room: initial mean arterial pressure (measured by the anesthesiologist), anesthesia technique, heavy bupivacaine spinal dose, Sufentanil spinal dose, fentanil spinal dose, morphine spinal dose, if received intravenous opioids, intraoperative nausea, intraoperative vomiting, lowest mean arterial pressure after anesthesia, if vasopressors were used and how (if prophylactic or after symptoms);
- 5. Some secondary outcome data will be collected in post anesthesia care unit (PACU) during the first 2 hours: nausea and intensity (0-10), vomiting episodes number.
- 6. The main outcome data will be collected 24 hours after the cesarean, for complications between 2-24 hours after the cesarean: nausea and intensity (0-10), vomiting episodes number.
- 7. Informed consent will be confirmed in the end by repeating explanations to the patient and asking her for signing the informed consent form.

Data will be collected electronically and a comma separated values file (CSV extension) will be generated for analysis. The file will be named NCT03171688.CSV